CLINICAL TRIAL: NCT07167966
Title: Alzheimer's Tau Platform (ATP): Regimen Specific Appendix for AADvac1
Brief Title: Alzheimer's Tau Platform: Regimen A - AADvac1
Acronym: ATP
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Paul S. Aisen (Other)
Collaborators: Axon Neuroscience SE (Industry); University of California, San Francisco (Other); Massachusetts General Hospital (Other); Alzheimer's Therapeutic Research Institute (Other); Alzheimer's Clinical Trials Consortium (Other); National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor-Investigator, Paul S. Aisen, Director, ATRI, University of Southern California
Organization: University of Southern California (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ATRI-014-A; R01AG078457 (NIH)
Record Dates: First submitted 2025-08-27; First posted 2025-09-11 (Actual); Last update posted 2025-09-26 (Actual); Status verified 2025-09

CONDITIONS: Preclinical Alzheimer's Disease; Prodromal Alzheimer's Disease; Alzheimer Disease
Keywords: anti-amyloid mAb; monoclonal antibody (mAB); tau; amyloid
MeSH Terms: conditions — Alzheimer Disease; Pick Disease of the Brain | interventions — AADvac1

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- AADvac1 monotherapy (Experimental): Intravenous infusions of anti-amyloid mAb-matched placebo for 6 months, followed by subcutaneous injections of AADvac1 over 24 months (n = 150)
  Interventions: Drug: AADvac1
- Combination AADvac1 therapy with anti-amyloid monoclonal antibody (mAb) (Experimental): Intravenous infusions of an anti-amyloid mAb for 6 months, combination anti-amyloid mAb and subcutaneous injections of AADvac1 for 6 months, followed by 18 months of AADvac1 injections alone (n = 150)
  Interventions: Drug: AADvac1; Drug: Anti-amyloid Monoclonal Antibody (mAb)
- Anti-amyloid monoclonal antibody (mAb) active control (Active Comparator): Intravenous infusions of an anti-amyloid mAb for 6 months, combination anti-amyloid mAb and AADvac1-matched placebo subcutaneous injections for 6 months, followed by 18 months of AADvac1-matched placebo injections alone (n = 75).
  Interventions: Drug: Anti-amyloid Monoclonal Antibody (mAb)

INTERVENTIONS:
Drug: AADvac1 — Subcutaneous injection of AADvac1
  Arms: AADvac1 monotherapy; Combination AADvac1 therapy with anti-amyloid monoclonal antibody (mAb)
Drug: Anti-amyloid Monoclonal Antibody (mAb) — Active comparator: intravenous infusion of an anti-amyloid mAb
  Arms: Anti-amyloid monoclonal antibody (mAb) active control; Combination AADvac1 therapy with anti-amyloid monoclonal antibody (mAb)

SUMMARY:
The Alzheimer's Tau Platform (ATP) is a multi-center platform trial to evaluate the safety and effectiveness of tau-directed therapies, alone or in combination with an anti-amyloid monoclonal antibody (mAb), in adults aged 50-80 with late preclinical or early prodromal Alzheimer's disease.

Regimen A will evaluate the safety and efficacy of AADvac1, alone or in combination with an anti-amyloid mAb.

DETAILED DESCRIPTION:
The Alzheimer's Tau Platform (ATP) is a multi-center platform trial to evaluate the safety and effectiveness of tau-directed therapies, alone or in combination with an anti-amyloid mAb, in adults aged 50-80 with late preclinical or early prodromal Alzheimer's disease. This platform trial allows for the simultaneous testing of multiple tau therapies under a shared master protocol. This means that multiple investigational products will be tested simultaneously or sequentially. Each investigational product will be tested in a regimen. The ATP Master Protocol is registered as NCT06957418.

Once a participant enrolls into the Master Protocol and meets all eligibility criteria, the participant will be eligible to be randomized into a currently enrolling regimen. All participants will have an equal chance of being randomized to any currently enrolling regimen.

Participants randomized to Regimen A - AADvac1 will be randomized in a 2:2:1 ratio to either AADvac1 alone, combination AADvac1 therapy with an anti-amyloid mAb, or an anti-amyloid mAb active control. The allocation ratio may be change based on the number of concurrent active regimens to ensure appropriate number of individuals randomized to the control arm across all active regimes.

Regimen A will enroll by invitation, as participants may not choose to enroll in a given regimen. Participants must first enroll into the Master Protocol and be eligible to participate in the Master Protocol before being able to be randomly assigned to Regimen A.

For a list of enrolling sites, please see the ATP Master Protocol under NCT06957418.

ELIGIBILITY:
Inclusion Criteria:

* No additional inclusion criteria beyond the inclusion criteria specified in the Master Protocol (NCT06957418).

Exclusion Criteria:

* No additional exclusion criteria beyond the exclusion criteria specified in the Master Protocol (NCT06957418).

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 375 (Estimated)
Dates: Start 2025-11 (Estimated); Primary Completion 2028-08-31 (Estimated); Study Completion 2028-08-31 (Estimated)

PRIMARY OUTCOMES:
Reduction of brain tau deposition as measured by tau positron emission tomography (PET) | 0, 6, 18 and 30 months
  To determine whether at least one tau therapy, either alone or in combination with an anti-amyloid mAb, will produce a greater reduction in brain tau deposition as measured by 18F-MK-6240 PET compared to anti-amyloid mAb alone.

SECONDARY OUTCOMES:
Disease progression as measured by plasma biomarkers | 30 months
  To assess whether at least one tau therapy, either alone or in combination with an anti-amyloid mAb slows disease progression as measured by plasma biomarkers.

CONTACTS AND LOCATIONS:
Overall Officials: Adam Boxer, MD, PhD, Principal Investigator — University of California, San Francisco (UCSF), Memory and Aging Center; Keith Johnson, MD, Principal Investigator — Massachusetts General Hospital (MGH), Harvard Medical School

IPD SHARING:
Plan to Share IPD: Yes